CLINICAL TRIAL: NCT00088673
Title: A Phase III Study of the Efficacy and Safety of 3APS in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Evaluation of 3APS in Patients With Mild to Moderate Alzheimer's Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-758007
Record Dates: First submitted 2004-07-30; First posted 2004-08-03 (Estimated); Last update posted 2007-02-28 (Estimated); Status verified 2007-02

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 3APS

SUMMARY:
The purpose of this Phase III study is to evaluate the efficacy and safety of 3APS compared to placebo (inactive substance pill) in patients with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in this study if they meet all of the following criteria:

* Male or Female (age 50 years and older): Female must be of non-childbearing potential (i.e. surgically sterilized or at least 2 years post-menopausal).
* Diagnosis of probable Alzheimer's disease based on the National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA criteria).
* Severity of dementia of mild to moderate degree as assessed by the Mini Mental State Examination (MMSE) performed at the screening visit.
* Patient must be living in the community with a reliable caregiver. Participant living in an assisted living facility may be included if study medication intake is supervised and participant has a reliable caregiver.
* Potential participant must be treated with conventional Alzheimer's disease therapies and must be on stable dose for at least 4 months prior to the screening visit and during the entire study period.
* Fluency in English, French or Spanish (oral and written).
* Signed informed consent from potential participant or legal representative and caregiver.

Exclusion Criteria:

Patients will not be eligible to participate in the study if they meet any of the following criteria:

* Potential participant with any other cause of dementia.
* Life expectancy less than 2 years.
* Potential participant with a clinically significant and/or uncontrolled condition or other significant medical disease.
* Use of an investigational drug within 30 days prior to the screening visit or during the entire study.
* Previous use of 3APS.

Patient recruitment is done by participating centers.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 950
Dates: Start 2004-06

PRIMARY OUTCOMES:
The two primary efficacy parameters are the change from baseline to month 18 in the Alzheimer's Disease Assessment Scale, cognitive subpart (ADAS-cog) and the clinical Deterioration Scale Sum of Boxes (CDR-SB) scores.
The brain volume change from baseline as measured by Magnetic Resonance Imaging will also be assessed.

CONTACTS AND LOCATIONS:
Locations (67):
- United States (50):
  - Pivotal Research Centers, Peoria, Arizona
  - 21st Century Neurology, a division of Xenoscience, Phoenix, Arizona
  - Central Arkansas Research, Hot Springs, Arkansas
  - Margolin Brain Institute, Fresno, California
  - Senior Clinical Trials, Inc., Laguna Hills, California
  - Pacific Research Network, Inc., San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Radiant Research, Denver, Colorado
  - Research Center for Clinical Studies, Inc., Darien, Connecticut
  - Yale University, Alzheimer's Disesase Research Unit, New Haven, Connecticut
  - New England Research Institute, Stamford, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Neuropsychiatric Research Center of SouthWest Florida, Fort Myers, Florida
  - Berma Research Group, Hialeah, Florida
  - Tukoi Institute for Clinical Research, Miami, Florida
  - Palm Beach Neurological Center, Palm Beach Gardens, Florida
  - Quantum Laboratories Inc at the Memory Disorders Clinic, North Broward Medical Center, Pompano Beach, Florida
  - Axiom Clinical Research, Tampa, Florida
  - Byrd Alzheimer's Center and Research Institute, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - University of South Florida, Suncoast Gerontology Center, Tampa, Florida
  - Premiere Research Institute Palm Beach Neurology, West Palm Beach, Florida
  - Comprehensive Neurology Specialists, PC, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Southern Illinois University (SIU) School of Medicine, Department of Neurology, Springfield, Illinois
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Mood & Memory Clinic - Dr Aronson, Farmington Hills, Michigan
  - Memory Enhancement Center, Long Branch, New Jersey
  - Neurological Associates of Albany, Albany, New York
  - Eastside Comprehensive Medical Center, New York, New York
  - NYU School of Medicine, New York, New York
  - Global Research and Consulting, Olean, New York
  - Nathan S. Kline Institute, Orangeburg, New York
  - University of Rochester-Program in Neurobehavioral Therapeutics, Rochester, New York
  - Richard H. Weisler, MD, PA and Associates, Raleigh, North Carolina
  - Wake Forest University School of Medicine, Department of Psychiatry and Behavioral Medicine, Winston-Salem, North Carolina
  - University Memory and Aging Center, Cleveland, Ohio
  - Neurology and Neuroscience Center of Ohio, Toledo, Ohio
  - Clinical Pharmaceuticals Trials, Inc., Tulsa, Oklahoma
  - CNS Research Institute, Philadelphia, Pennsylvania
  - Farber Institute for Neurosciences, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh ADRC, Pittsburgh, Pennsylvania
  - CNS Research, Inc., East Providence, Rhode Island
  - Memory and Aging Program, Butler Hospital, Providence, Rhode Island
  - MUSC - Alzheimer's Research and Clinical Programs, North Charleston, South Carolina
  - Clinical Research Services at Tennessee Christian Medical Center, Madison, Tennessee
  - University of Texas Mental Sciences Institute, Houston, Texas
  - Air Force Villages-Freedom House Research (Study open to Air Force Village residents only), San Antonio, Texas
  - The Memory Clinic, Bennington, Vermont
- Canada (17):
  - Calgary, Alberta
  - The Medical Arts Health Research Group, a Division of PCT Networks, Inc., Penticton, British Columbia
  - St. Joseph's Hospital, Saint John, New Brunswick
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Queen's University, Kingston, Ontario
  - Geriatric Clinical Trials Group, Parkwood Hospital, London, Ontario
  - Ottawa, Ontario
  - Gerontion Research, Toronto, Ontario
  - Sunnybrook and Women's College Health Science Centre, Toronto, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Clinique Neuro Rive-Sud, Greenfield Park, Quebec
  - Hôpital Maisonneuve-Rosemont, Recherche Clinique de Neurologie, Montreal, Quebec
  - Jewish General Hospital- Memory Clinic, Montreal, Quebec
  - Hôpital de l'Enfant-Jésus, Québec, Quebec
  - Memory & Motor Skills Disorders Clinic, Québec, Quebec
  - Centre de recherche Novabyss, Sherbrooke, Quebec
  - McGill Centre for Studies in Aging, Verdun (Montreal), Quebec